CLINICAL TRIAL: NCT02825082
Title: Risk Stratification Tools and Frailty Index for Predicting Perioperative Outcome in Elderly Patients Undergoing Abdominal Emergency Surgery
Brief Title: Emergency Surgery in the Elderly: Comparison of Frailty Index and Surgical Risk Score
Acronym: FRAILESEL
Status: Completed | Type: Observational
Sponsor: University of Roma La Sapienza (Other)
Responsible Party: Principal Investigator, Gianluca Costa, MD, PhD,, University of Roma La Sapienza
Other Study IDs: 4252_2016 - 12/12/2016
Record Dates: First submitted 2016-06-28; First posted 2016-07-07 (Estimated); Last update posted 2018-08-28 (Actual); Status verified 2018-08

CONDITIONS: Surgery; Emergency
Keywords: Emergency general surgery; Geriatric; Outcomes; Frailty
MeSH Terms: conditions — Emergencies; Frailty

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Abdominal emergency surgery — all abdominal emergency surgery procedures

SUMMARY:
EMERGENCY GENERAL SURGERY IN GERIATRIC PATIENTS: EPIDEMIOLOGY, AND EVALUATION OF FACTORS AFFECTING MORBIDITY AND MORTALITY

DETAILED DESCRIPTION:
BACKGROUND: nowadays becoming old is considered a results from the socioeconomic development and improvements in health care systems worldwide. The life expectancy of the average person doubled over the course of the last century and it is currently estimated at 85-90 years in western countries.. The number of elderly people will increase dramatically over the next few decades with population projections towards 2040 indicating a 66% increase in the age-groups 65 to 74 years. More importantly, the age groups 75 years and above are projected to increase with >100%, which clearly will have implications for future health services. Thus, an acute medical insult may thus deprive a healthy 65- or 75-years old person from a considerable numbers of future life-years (20-30 years), either as lived in dependency. Older adults make up a large portion of surgical practice worldwide. In 2010, 37% of all inpatient operations performed in the United States were in patients 65 years and older, and this percentage will rise in the coming decades. Also, with increasing age comes an added risk of additional disease as well as the use of drugs, some of which clearly can interfere with emergency surgical conditions. Elderly patients with life-threatening abdominal disease are undergoing emergency surgery in increasing numbers and despite recent advances in surgical and anaesthetic techniques, elderly patients are at increased risk for major perioperative complications such as delirium, urinary incontinence, pressure ulcers,depression, infection, functional decline and adverse drug affects, longer hospital stays, and postoperative institutionalization. Even after controlling for co-morbid illnesses and functional impairment, age remains an independent risk factor for adverse postoperative events. Elderly who receive acute surgery often survives the initial treatment, but often suffers from severe complications due to comorbidity. If a complication occurs, it can lead to a cascade of events resulting in disability, loss of independence, diminished quality of life, high health care costs, and mortality. It is important with close post-operative follow up to avoid life threatening complicating conditions, and to involve geriatric consultants and other specialties if needed. Additional surgery and aggressive life-prolonging care, can in some cases, do more harm than good. Surgical decision making in this population is challenging because of the heterogeneity of health status in older adults and the paucity of tools for predicting operative risk. Commonly used predictors of postoperative complications have substantial limitations; most are based on a single organ system or are subjective, and none estimate a patient's physiologic reserves. therefore may need to undergo special pretreatment assessments that incorporate frailty assessments. Frailty is commonly associated with older adults and is identified by decreased reserves in multiple organ systems because of disease, lack of activity, inadequate nutrition, stress, and the physiological changes of aging. Given the inevitable rise of the aging population, it is vital that surgeons understand the concept of frailty and how it may affect surgical decisions and outcomes. Improving outcomes in emergency surgery for the geriatric population is a multifaceted task but has great clinical and health care system implications. valuation of current practice is important to improve outcomes for the future. Acting on the identified deficits and finding new areas for research is important to improve outcomes in the elderly.

AIM: to evaluate stratification of the surgical risk in patient > 65yo underwent general emergency surgery. To evaluate specific parameters as variables for new score in the elderly patient. To underline hotspot in the managements of such patients.

STUDY DESIGN: both retrospective and prospective cohort, multicenter, observational, no profit clinical study. All the study participants will collect data on elderly patients underwent general emergency surgery during a 18 month old period, guaranteeing a whole completeness of the picked data > 95%. This study was approved by the Health Sciences Research Ethics Board of the University of Rome La Sapienza.

ELIGIBILITY:
Inclusion Criteria: All elderly patients submitted to emergency surgery considered as not-scheduled procedure within 7 days from admission

Exclusion Criteria: None

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Multicenter italian national survey cohort study
Sampling Method: Non-Probability Sample
Enrollment: 2200 (Actual)
Dates: Start 2017-01; Primary Completion 2017-12 (Actual); Study Completion 2018-06 (Actual)

PRIMARY OUTCOMES:
30-day mortality rate | 18 months
30-day morbidity rate | 18 months
  Morbidity defined by mean of the Clavien's Classification scoring system

SECONDARY OUTCOMES:
Portsmouth-Physiological and Operative Severity Score for the enumeration of Mortality and morbidity (P-POSSUM) | 18 months
  Observed to expected (O:E) mortality ratio
Calculation of Charlson Age-Comorbidity Index (CACI) | 18 months
  Calculation and evaluation of its predictive value for morbidity and mortality
Simplified Acute Physiology Score-II (SAPS-II) | 18 months
  Calculation and evaluation of its predictive value for mortality
American College of Surgeons National Surgical Quality Improvement Program (ACS NSQIP) surgical risk calculator | 18 months
  Calculation and evaluation of its predictive value for post-operative complications
Calculation of post-Operative Risk in Emergency Surgery (CORES) | 18 months
  Calculation and evaluation of its predictive value for mortality
Surgical mortality probability model (S-MPM) | 18 months
  Observed to expected (O:E) mortality ratio
Colorectal-Physiological and Operative Severity Score for the enumeration of Mortality and morbidity (CR-POSSUM) | 18 months
  Observed to expected (O:E) mortality ratio
Frailty Fried Index | 18 months
  Frailty stratification in participants
Canadian Study of Health and Ageing (CSHA) frailty score | 18 months
  Frailty stratification in participants
Total number of subjects underwent emergency surgery | 18 months
  Elderly to non elderly patient ratio
Geographical area inhabitants | 18 months
  Emergency surgery in the elderly per 100.000 inhabitants

CONTACTS AND LOCATIONS:
Overall Officials: Gianluca Costa, MD, PhD, Study Director — University of Roma La Sapienza, Sant' Andrea University Hospital; Giuseppe Nigri, MD, FACS, Principal Investigator — University of Roma La Sapienza, Sant' Andrea University Hospital
Locations (43):
- Italy (43):
  - Ospedale Civile Spirito Santo, Pescara, Abruzzo
  - Azienda Ospedaliero-Universitaria Consorziale Policlinico di Bari, Bari, Apulia
  - Presidio Ospedaliero Centrale SS Annunziata di Taranto, Taranto, Apulia
  - Policlinico San Pietro, Ponte San Pietro, Bergamo
  - Presidio Ospedaliero Duilio Casula, Monserrato, Cagliari, Sardegna
  - Ospedale Convenzionato Villa dei Fiori, Acerra, Campania
  - Azienda Ospedaliera di Rilievo Nazionale e di alta Specialità, Avellino, Campania
  - A.O.R.N Gaetano Rummo, Benevento, Campania
  - Azienda Ospedaliera Cardarelli, Napoli, Campania
  - Ospedale M. Bufalini Cesena, Cesena, Emilia-Romagna
  - Arcispedale S. Anna di Cona - Azienda Ospedaliero-Universitaria di Ferrara, Ferrara, Emilia-Romagna
  - Ospedale Maggiore di Parma, Parma, Emilia-Romagna
  - Ospedale Infermi, Rimini, Emilia-Romagna
  - Ospedale del Delta, Lagosanto, Ferrara
  - AAS2 Bassa Friulana Isotina - Presidio Ospedaliero di Gorizia, Monfalcone, Gorizia
  - Presidio Ospedaliero San Filippo Neri, Rome, Lazio
  - Azienda Ospedaliera San Camillo Forlanini di Roma, Rome, Lazio
  - Ospedale Cristo Re, Rome, Lazio
  - Policlinico Umberto I, Rome, Lazio
  - Ospedale Papa Giovanni XXIII, Bergamo, Lombardy
  - Fondazione IRCCS Ca' Granda - Ospedale Maggiore Policlinico, Milan, Lombardy
  - Ospedale Civile Sant'Agostino Estense, Baggiovara, Modena
  - Ospedale Civile di Voghera, Voghera, Pavia
  - Azienda Ospedaliero-Universitaria città della salute e della scienza di Torino, presidio Molinette, Turin, Piedmont
  - Ospedale Civile di Adria, Adria, Rovigo
  - Azienda Ospedaliera G. Brotzu, Cagliari, Sardinia
  - P.O. Santissima Trinità ASL8, Cagliari, Sardinia
  - Ospedale San Francesco, Nuoro, Sardinia
  - Ospedale Santissima Annunziata A.O.U. Sassari, Sassari, Sardinia
  - Azienda Ospedaliero-Universitaria Policlinico Vittorio Emanuele, Catania, Sicily
  - Azienda Ospedaliero Universitaria Ospedale Riuniti Ancona, Ancona, The Marches
  - Ospedale San Donato, Arezzo, Tuscany
  - Ospedale della Misericordia Grosseto, Grosseto, Tuscany
  - Azienda Ospedaliera Pisana Policlinico Universitario Cisanello, Pisa, Tuscany
  - Ospedale San Jacopo di Pistoia, Pistoia, Tuscany
  - Ospedale San Giovanni Battista, Foligno, Umbria
  - Ospedale Santa Maria della Stella, Orvieto, Umbria
  - Azienda Ospedaliera Santa Maria, Terni, Umbria
  - Policlinico Abano Terme, Abano Terme, Veneto
  - ULSS21 Legnago (Verona_ASL2), Legnago, Verona
  - Ospedale di Civita Castellana, Civita Castellana, Viterbo
  - Ospedale di Macerata, Marche
  - Azienda Ospedaliera Universitaria Policlinico Paolo Giaccone, Palermo

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] A, Frezza B, Scandavini CM, Fransvea P, Costa G, Balducci Mortalità e morbilità per chirurgia colica in urgenza nel paziente anziano Lo Conte G Osp. Ital. Chirurgia 2012
- [Background] Costa G, Nigri G, Tierno SM, Tomassini F, Varano GM, Venturini Emergency abdominal surgery in the elderly: a ten-year experience L BMC Geriatrics 2009, 9(Suppl 1):A53
- [Result] Joseph B, Zangbar B, Pandit V, Fain M, Mohler MJ, Kulvatunyou N, Jokar TO, O'Keeffe T, Friese RS, Rhee P. Emergency General Surgery in the Elderly: Too Old or Too Frail? J Am Coll Surg. 2016 May;222(5):805-13. doi: 10.1016/j.jamcollsurg.2016.01.063. Epub 2016 Feb 26. PMID 27113515
- [Result] Shah AA, Zafar SN, Kodadek LM, Zogg CK, Chapital AB, Iqbal A, Greene WR, Cornwell EE 3rd, Havens J, Nitzschke S, Cooper Z, Salim A, Haider AH. Never giving up: outcomes and presentation of emergency general surgery in geriatric octogenarian and nonagenarian patients. Am J Surg. 2016 Aug;212(2):211-220.e3. doi: 10.1016/j.amjsurg.2016.01.021. Epub 2016 Mar 19. PMID 27086200
- [Result] Hewitt J, McCormack C, Tay HS, Greig M, Law J, Tay A, Asnan NH, Carter B, Myint PK, Pearce L, Moug SJ, McCarthy K, Stechman MJ. Prevalence of multimorbidity and its association with outcomes in older emergency general surgical patients: an observational study. BMJ Open. 2016 Mar 31;6(3):e010126. doi: 10.1136/bmjopen-2015-010126. PMID 27033960
- [Result] Poldermans D, Hoeks SE, Feringa HH. Pre-operative risk assessment and risk reduction before surgery. J Am Coll Cardiol. 2008 May 20;51(20):1913-24. doi: 10.1016/j.jacc.2008.03.005. PMID 18482658
- [Result] Vasivej T, Sathirapanya P, Kongkamol C. Incidence and Risk Factors of Perioperative Stroke in Noncardiac, and Nonaortic and Its Major Branches Surgery. J Stroke Cerebrovasc Dis. 2016 May;25(5):1172-1176. doi: 10.1016/j.jstrokecerebrovasdis.2016.01.051. Epub 2016 Feb 24. PMID 26922129
- [Result] McLean RC, McCallum IJ, Dixon S, O'Loughlin P. A 15-year retrospective analysis of the epidemiology and outcomes for elderly emergency general surgical admissions in the North East of England: A case for multidisciplinary geriatric input. Int J Surg. 2016 Apr;28:13-21. doi: 10.1016/j.ijsu.2016.02.044. Epub 2016 Feb 23. PMID 26892599
- [Result] Merani S, Payne J, Padwal RS, Hudson D, Widder SL, Khadaroo RG. Predictors of in-hospital mortality and complications in very elderly patients undergoing emergency surgery. World J Emerg Surg. 2014 Jul 7;9:43. doi: 10.1186/1749-7922-9-43. eCollection 2014. PMID 25050133
- [Result] Desserud KF, Veen T, Soreide K. Emergency general surgery in the geriatric patient. Br J Surg. 2016 Jan;103(2):e52-61. doi: 10.1002/bjs.10044. Epub 2015 Dec 1. PMID 26620724
- [Result] St-Louis E, Sudarshan M, Al-Habboubi M, El-Husseini Hassan M, Deckelbaum DL, Razek TS, Feldman LS, Khwaja K. The outcomes of the elderly in acute care general surgery. Eur J Trauma Emerg Surg. 2016 Feb;42(1):107-13. doi: 10.1007/s00068-015-0517-9. Epub 2015 Apr 8. PMID 26038035
- [Result] Lorenzon L, Costa G, Massa G, Frezza B, Stella F, Balducci G. The impact of frailty syndrome and risk scores on emergency cholecystectomy patients. Surg Today. 2017 Jan;47(1):74-83. doi: 10.1007/s00595-016-1361-1. Epub 2016 May 30. PMID 27241560
- [Result] Costa G, La Torre M, Frezza B, Fransvea P, Tomassini F, Ziparo V, Balducci G. Changes in the surgical approach to colonic emergencies during a 15-year period. Dig Surg. 2014;31(3):197-203. doi: 10.1159/000365254. Epub 2014 Aug 28. PMID 25170867
- [Result] Costa G, Tomassini F, Tierno SM, Venturini L, Frezza B, Cancrini G, Mero A, Lepre L. [Emergency colonic surgery: analysis of risk factors predicting morbidity and mortality]. Chir Ital. 2009 Sep-Dec;61(5-6):565-71. Italian. PMID 20380259
- [Derived] Costa G, Massa G; ERASO (Elderly Risk Assessment for Surgical Outcome) Collaborative Study Group. Frailty and emergency surgery in the elderly: protocol of a prospective, multicenter study in Italy for evaluating perioperative outcome (The FRAILESEL Study). Updates Surg. 2018 Mar;70(1):97-104. doi: 10.1007/s13304-018-0511-y. Epub 2018 Jan 30. PMID 29383680